CLINICAL TRIAL: NCT05895422
Title: Functional Outcome After Laparoscopic and Robot Assisted Management of Uretero-pelvic Junction Obstruction Disease Caused by Crossing Vessels for Adult Patients
Brief Title: Functional Outcome After Minimally Invasive Pyeloplasty for Adult Patients With UPJO
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Rammah, lecturer of urology- faculty of medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MD-85-2023
Record Dates: First submitted 2023-05-31; First posted 2023-06-08 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Ureteropelvic Junction Obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral

STUDY DESIGN:
Intervention Model Description: randomized intervention study
Who Masked: Participant
Masking Description: one blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vascular hitch (Experimental): displacement of the lower polar crossing vessels causing the UPJO
  Interventions: Procedure: pyeloplasty
- Dismembered pyeloplasty (Active Comparator): classic Anderson-Hynes procedure
  Interventions: Procedure: pyeloplasty

INTERVENTIONS:
Procedure: pyeloplasty — repair of the uPJO

SUMMARY:
an intervention study on adult patients with uretero-pelvic junction obstruction (UPJO) due to crossing vessels would be managed either through classic dismembered pyeloplasty or vascular hitch.

DETAILED DESCRIPTION:
in recent studies, some patients with crossing vessels UPJO could be managed by vascular displacement of these vessels, what is named as vascular hitch or vasculopexy in a way to avoid classic dismembered technique. this newer technique is supposed to provide comparable results to the classic technique but with lesser operative time and shorter hospital stay. in the era of minimally invasive procedures, robotic assisted or laparoscopic vascular hitch could provide many advantages over the classic open technique.

ELIGIBILITY:
Inclusion Criteria:

* all patients with UPJO above 18 years
* UPJO caused by crossing vessels confirmed by CT angiography
* Symptomatic UPJO

Exclusion Criteria:

* recurrent UPJO after a previous trial of open repair ,
* secondary UPJO after open renal surgery.
* UPJO in non functioning kidney

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
comparing the two techniques regarding the success rate | 2 years
  both techniques are supposed to have similar results

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
the researchers would determine whether they would share or not during the study